CLINICAL TRIAL: NCT01920685
Title: Computerised Interventions for Thinking and Anxiety in Delusions (CITADEL) Trial
Acronym: CITADEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Amy Hardy, Research Clinical Psychologist, King's College London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13/LO/0690
Record Dates: First submitted 2013-08-05; First posted 2013-08-12 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Paranoia in People With Schizophrenia-spectrum Diagnosis
Keywords: Paranoia; CBT; Reasoning; Anxiety
MeSH Terms: conditions — Paranoid Disorders; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate therapy (Experimental): 6 sessions of talking therapy, targeting anxiety processes associated with paranoia, will be delivered for a period of 8 weeks immediately after randomisation.
  Interventions: Other: Anxiety intervention
- Delayed intervention (Other): Therapy will be delayed until 12 weeks following randomisation, and then 6 sessions of talking therapy, targeting anxiety processes associated with paranoia, will be delivered over a period of 8 weeks.
  Interventions: Other: Anxiety intervention

INTERVENTIONS:
Other: Anxiety intervention

SUMMARY:
People with a schizophrenia spectrum diagnosis often experience distressing worries or beliefs about others intending to cause them harm (also known as paranoia). Paranoid beliefs are associated with significant distress and disruption to the person's life. This results in high use of services and costs to mental health providers.

The National Institute of Clinical Excellence recommends that cognitive behavioural therapy for psychosis (CBTp) is offered to everybody with a schizophrenia spectrum psychosis. The latest meta analyses report improved outcomes, and reduced inpatient stays following CBTp, making it a cost effective intervention.

Although improved outcomes have been obtained by therapies, CBTp has only small to moderate effects on paranoid beliefs. Further, training therapists to competently deliver CBTp is intensive, expensive and takes up to a year. CBTp is therefore not widely available to service users, resulting in inequalities in access to care.

The investigators are seeking to improve outcomes and accessibility of CBTp for people with distressing, paranoid beliefs. The proposed research programme aims to conduct a feasibility study of a brief therapeutic intervention, aimed at targeting and improving anxiety processes that are causally implicated in paranoia (Freeman et al, 2015).

The investigators have preliminary evidence indicating that the pilot intervention, with interactive multimedia content, reduced distressing beliefs and improved coping (Freeman et al, 2015). Participants also reported they found the therapy acceptable, enjoyable and useful. Based on these results, the investigators have further modified the intervention. The feasibility and efficacy of the therapy will be investigated in a randomised controlled design (n = 34).

Please note the protocol has been been amended to exclude a pilot trial of a second brief intervention targeting reasoning styles in paranoia, as since the initial protocol was developed we have obtained data from two randomised pilot studies demonstrating its feasibility and acceptability (Garety et al, 2015; Waller et al, 2015). A further pilot trial of the reasoning styles intervention is therefore not indicated.

ELIGIBILITY:
Inclusion Criteria:

* Self reported worries about being harmed or at risk from others
* Non-affective psychosis(ICD10,F20-F29)
* Age 18-65
* Symptoms stable no major relapse or crisis in last 3 months prior to consent
* Sufficient command of English to provide informed consent, complete the measures and participate in the brief interventions
* Score above the cutoff for clinically significant levels of paranoia on the Green Paranoid Thoughts Scale (Green et al, 2008)
* Paranoia is triggered by being outside

Exclusion Criteria:

* Lack of capacity to provide informed consent
* Primary diagnosis of drug or alcohol use with secondary psychosis
* Primary diagnosis of mood disorder or bipolar affective disorder
* Primary diagnosis of learning difficulty
* Unstable residential arrangements (making a move away during the course of participation in the research likely)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Green Paranoid Thoughts Scale | Change from baseline in paranoia scores at 8 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Garety, CPsychol, MPhil, PhD, FBPsS, Study Chair — King's College London
Locations (2):
- United Kingdom (2):
  - Oxleas NHS Foundation Trust, Dartford, Kent
  - South London & Maudsley NHS Foundation Trust, London, London

REFERENCES:
- [Background] Freeman D, Emsley R, Dunn G, Fowler D, Bebbington P, Kuipers E, Jolley S, Waller H, Hardy A, Garety P. The Stress of the Street for Patients With Persecutory Delusions: A Test of the Symptomatic and Psychological Effects of Going Outside Into a Busy Urban Area. Schizophr Bull. 2015 Jul;41(4):971-9. doi: 10.1093/schbul/sbu173. Epub 2014 Dec 20. PMID 25528759
- [Background] Freeman D, Waller H, Harpur-Lewis RA, Moore R, Garety P, Bebbington P, Kuipers E, Emsley R, Dunn G, Fowler D, Jolley S. Urbanicity, persecutory delusions, and clinical intervention: the development of a brief CBT module for helping patients with persecutory delusions enter social urban environments. Behav Cogn Psychother. 2015 Jan;43(1):42-51. doi: 10.1017/S1352465813000660. Epub 2013 Aug 9. PMID 23930939
- [Background] Garety P, Waller H, Emsley R, Jolley S, Kuipers E, Bebbington P, Dunn G, Fowler D, Hardy A, Freeman D. Cognitive mechanisms of change in delusions: an experimental investigation targeting reasoning to effect change in paranoia. Schizophr Bull. 2015 Mar;41(2):400-10. doi: 10.1093/schbul/sbu103. Epub 2014 Jul 21. PMID 25053650
- [Background] Waller H, Emsley R, Freeman D, Bebbington P, Dunn G, Fowler D, Hardy A, Kuipers E, Garety P. Thinking Well: A randomised controlled feasibility study of a new CBT therapy targeting reasoning biases in people with distressing persecutory delusional beliefs. J Behav Ther Exp Psychiatry. 2015 Sep;48:82-9. doi: 10.1016/j.jbtep.2015.02.007. Epub 2015 Feb 24. PMID 25770671